CLINICAL TRIAL: NCT03524703
Title: Short-term Effect of Chewing Gum in Patients With Mild-moderate Dysphagia After Anterior Cervical Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, YunBing Chang, Head of Spine Department, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GDREC 2018151H
Record Dates: First submitted 2018-04-11; First posted 2018-05-15 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Dysphagia
Keywords: dysphagia; anterior cervical fusion; chewing gum
MeSH Terms: conditions — Deglutition Disorders | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing Gum Group (Experimental): Patients who receive anterior cervical fusion and have mild or moderate dysphagia postoperatively, will be randomized into two groups. Subjects assigned to the Chewing Gum Group are asked to chew gum four times a day for 5 days (15 minutes each time) after surgery in addition to standard cares. Standard cares include cleaning the wound every 2 days, wearing a collar, pain management, and education.
  Interventions: Other: chewing gum
- Control Group (No Intervention): Patients who receive anterior cervical fusion and have mild or moderate dysphagia postoperatively, will be randomized into two groups. Subjects assigned to the Control Group receive standard cares and are asked not to chew gum within 5 days after surgery. Standard cares include cleaning the wound every 2 days, wearing a collar, pain management, and education.

INTERVENTIONS:
Other: chewing gum — Chewing gum four times per day for 5 days, 15 minutes each time.
  Arms: Chewing Gum Group

SUMMARY:
The aim of the study is to estimate the effect of chewing gum after anterior cervical fusion surgery on decreasing the severity of dysphagia in patients with mild-moderate dysphagia.

DETAILED DESCRIPTION:
Postoperative dysphagia is the most common complication of anterior cervical fusion surgery. Previous studies showed that chewing gum helped to improve swallow frequency and latency. However, its short-term effect on alleviating dysphagia symptom after anterior cervical surgery is still unknown. A randomized, parallel controlled, superiority trial is performed in patients with postoperative mild-moderate dysphagia. Dysphagia severity will be assessed using dysphagia short questionnaire (DSQ) score in the chewing gum group and control group during 7 days after surgery, and the changes in DSQ score between two groups will be compared, to estimate the effect of chewing gum on alleviating dysphagia symptom.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 years to 80 years.
* underwent anterior cervical fusion surgery for degenerative cervical disease.
* diagnosed with mild or moderate postoperative dysphagia 1 day after surgery using Bazaz scale.

Exclusion Criteria:

* Patients underwent revision procedures or procedures treating conditions other than degenerative cervical disease.
* Patients with preoperative dysphagia.
* Patients unable to chew, or unable to follow the directions for chewing gum.
* Patients unable to attend follow-up visits or finish the dysphagia questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-04-28 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Short Questionnaire (DSQ) score | Change from the 1st day after surgery to the 7th day after surgery.
  DSQ is designed for the evaluation of swallowing difficulty after anterior cervical spine surgery. It is calculated by summing up the points given for each item, from 0 point to a maximum of 18 points, where lower scores represent milder symptoms and vice versa.

SECONDARY OUTCOMES:
Bazaz grading system | Change from the 1st day after surgery to the 7th day after surgery.
  Bazaz grading system is designed for the evaluation of swallowing difficulty after anterior cervical spine surgery. The patients are graded as having none, mild, moderate, or severe dysphagia based on their symptoms. A none or mild dysphagia is considered to be a better outcome.
Prevertebral soft tissue swelling | The 3rd days after surgery.
  The measurement of the soft tissue space is made on the line parallel to the upper end plate from the midpoint of the anterior surface of each vertebral body to the border of the airway shadow. This scale ranges from 0 to approximately 30 mm for each vertebra, where a lower value represents a milder soft tissue swelling.

CONTACTS AND LOCATIONS:
Overall Officials: Yunbing Chang, M.D., Ph.D., Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT03524703/Prot_SAP_000.pdf